CLINICAL TRIAL: NCT05542784
Title: Modified Laparoendoscopic Rendezvous for Secondary Choledocholithiasis: a Nonrandomized Controlled Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20223357016
Record Dates: First submitted 2022-07-29; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-05

CONDITIONS: Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with choledocholithiasis secondary to choledocholithiasis undergoing LERV surgery
  Interventions: Procedure: Modified LERV
- Patients with choledocholithiasis secondary to choledocholithiasis undergoing PreERCP+LC surgery

INTERVENTIONS:
Procedure: Modified LERV — Patients routinely underwent LC. The ligature clamp clamps the distal end of the capsule tube. In this case, you need to perform two steps:
  Laparoscopic operation: proximal incision, anterograde placement of guide wire into the duodenum. The catheter was removed and the balloon dilated. The balloon was released and removed when the ERCP was initiated for cannulation. After successful ERCP retrograde placement, the anterograde guide wire was pulled out and the gallbladder was removed.
  ERCP procedure: After the anterograde guide wire was observed by duodenoscope, duodenal papilla was placed through a retrograde incision along the anterograde guide wire, and a retrograde cannula was inserted into the common bile duct. Remove stones by dragging them with a net basket or/and balloon. Angiography confirmed that there was no filling defect in the extrahepatic bile duct, and ENBD was indwelled.
  Other Names: Pre ERCP+LC
  Groups: Patients with choledocholithiasis secondary to choledocholithiasis undergoing LERV surgery

SUMMARY:
This study intends to explore the success rate and clinical efficacy of modified LERV in the treatment of patients with non-dilated common bile duct (internal diameter ≤10mm) through a non-randomized controlled clinical trial, and to clarify whether modified LERV can be used as the preferred routine treatment for choledocholithiasis secondary to gallbladder stones.

DETAILED DESCRIPTION:
Patients with cholecystolithiasis secondary to common bile duct stones requiring surgical treatment during a 3-year period from 2022-6-1 to 2025-3-31 were enrolled in this non-randomized controlled clinical trial. Preoperative diameter of the middle common bile duct was determined by magnetic resonance cholangiography (MRCP) or B-ultrasound measurement. The actual treatment plan of the patients was recorded, including LERV treatment and ERCP+LC treatment. The baseline data and the success rate of stone removal, operation time, postoperative stone residual rate, complication rate, length of hospital stay and hospitalization cost were recorded for observation and follow-up. To determine whether modified LERV can be used as the preferred routine treatment for choledocholithiasis secondary to gallbladder stones.

ELIGIBILITY:
Inclusion Criteria:

1、18 years ≤ age <85 years 2、clinical diagnosis of choledocholithiasis secondary to cholecystolithiasis and middle choledocholithiasis (MCBD) diameter ≤10mm; The diameter of MCBD was based on MRCP measurements. If MRCP could not be performed, CT images were used as reference, and B-ultrasound measurements were used as the standard.

3、 Good cardiopulmonary function, anesthesia evaluation tolerance under general anesthesia laparoscopic + endoscopic surgery.

-

Exclusion Criteria:

1、 Intrahepatic bile duct stones with indications for surgery, and need simultaneous surgery; 2、 Patients with choledocholithiasis >2 cm or a large number of stones were difficult to remove; 3、 Patients with malignant hepatobiliary and pancreatic tumors or biliary tract malformations; 4、 Severe patients with severe pancreatitis and septic shock before operation; 5、Patients with previous gastric and duodenoscopic surgery history and interruption of gastroduodenal continuity; 6、 Severe partial stenosis of the upper gastrointestinal tract (from the oral cavity to the second duodenum), which is expected to be inaccessible to the duodenoscope.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 85 years with common bile duct stones who are suitable for and consent to undergo laparoscopic plus endoscopic surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness evaluation index | intraoperative
  Success rate of stone removal (as judged by ERCP imaging)

SECONDARY OUTCOMES:
Postoperative related clinical indicators | Blood routine, pancreatic enzyme binomial and liver function were examined on the first and second day after operation.
  The incidence of PEP
The hospital indicators | an average 1 week
  Length of hospital stay after operation (including operation day), hospitalization cost after operation (including operation day)
the incidence of serious complications | Within 1 year
  including duodenal papilla hemorrhage, duodenal perforation, acute pancreatitis, duodenal leakage (fistula), abdominal abscess, the incidence of hyperamylasemia, the incidence of residual common bile duct stones, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zibing Fan, Attending physician, Study Chair — Shenzhen Second People's Hospital; Ganchen Sun, Nurse practitioner, Study Chair — Shenzhen Second People's Hospital; Yanan Bao, nurse-in-charge, Study Chair — Shenzhen Second People's Hospital; Xuelin Liu, Nurse practitioner, Study Chair — Shenzhen Second People's Hospital; Haoyuan Deng, Attending physician, Study Chair — Shenzhen Second People's Hospital; Yifan Zhang, Master's Degree student, Study Chair — Shenzhen Second People's Hospital; Yang Li, Nurse practitioner, Study Chair — Shenzhen Second People's Hospital; Haoran Ma, Nurse practitioner, Study Chair — Shenzhen Second People's Hospital; Naiyang Zhan, Attending physician, Study Chair — Shenzhen Second People's Hospital; Yiyuan Chen, Master's Degree student, Study Chair — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tazuma S. Gallstone disease: Epidemiology, pathogenesis, and classification of biliary stones (common bile duct and intrahepatic). Best Pract Res Clin Gastroenterol. 2006;20(6):1075-83. doi: 10.1016/j.bpg.2006.05.009. PMID 17127189
- [Result] Bradley A, Sami S, Hemadasa N, Macleod A, Brown LR, Apollos J. Decision analysis of minimally invasive management options for cholecysto-choledocholithiasis. Surg Endosc. 2020 Dec;34(12):5211-5222. doi: 10.1007/s00464-020-07816-w. Epub 2020 Jul 24. PMID 32710213
- [Result] Deslandres E, Gagner M, Pomp A, Rheault M, Leduc R, Clermont R, Gratton J, Bernard EJ. Intraoperative endoscopic sphincterotomy for common bile duct stones during laparoscopic cholecystectomy. Gastrointest Endosc. 1993 Jan-Feb;39(1):54-8. doi: 10.1016/s0016-5107(93)70011-5. No abstract available. PMID 8454146
- [Result] Liu W, Wang Q, Xiao J, Zhao L, Huang J, Tan Z, Li P. A modified technique reduced operative time of laparoendoscopic rendezvous endoscopic retrograde cholangiopancreatography combined with laparoscopic cholecystectomy for concomitant gallstone and common bile ductal stone. Gastroenterol Res Pract. 2014;2014:861295. doi: 10.1155/2014/861295. Epub 2014 Jun 15. PMID 25024701
- [Result] Mine T, Morizane T, Kawaguchi Y, Akashi R, Hanada K, Ito T, Kanno A, Kida M, Miyagawa H, Yamaguchi T, Mayumi T, Takeyama Y, Shimosegawa T. Clinical practice guideline for post-ERCP pancreatitis. J Gastroenterol. 2017 Sep;52(9):1013-1022. doi: 10.1007/s00535-017-1359-5. Epub 2017 Jun 26. PMID 28653082
- [Result] Bailey AA, Bourke MJ, Williams SJ, Walsh PR, Murray MA, Lee EY, Kwan V, Lynch PM. A prospective randomized trial of cannulation technique in ERCP: effects on technical success and post-ERCP pancreatitis. Endoscopy. 2008 Apr;40(4):296-301. doi: 10.1055/s-2007-995566. PMID 18389448
- [Result] Cotton PB, Garrow DA, Gallagher J, Romagnuolo J. Risk factors for complications after ERCP: a multivariate analysis of 11,497 procedures over 12 years. Gastrointest Endosc. 2009 Jul;70(1):80-8. doi: 10.1016/j.gie.2008.10.039. Epub 2009 Mar 14. PMID 19286178
- [Result] ASGE Standards of Practice Committee; Buxbaum JL, Abbas Fehmi SM, Sultan S, Fishman DS, Qumseya BJ, Cortessis VK, Schilperoort H, Kysh L, Matsuoka L, Yachimski P, Agrawal D, Gurudu SR, Jamil LH, Jue TL, Khashab MA, Law JK, Lee JK, Naveed M, Sawhney MS, Thosani N, Yang J, Wani SB. ASGE guideline on the role of endoscopy in the evaluation and management of choledocholithiasis. Gastrointest Endosc. 2019 Jun;89(6):1075-1105.e15. doi: 10.1016/j.gie.2018.10.001. Epub 2019 Apr 9. PMID 30979521
- [Result] Noel R, Enochsson L, Swahn F, Lohr M, Nilsson M, Permert J, Arnelo U. A 10-year study of rendezvous intraoperative endoscopic retrograde cholangiography during cholecystectomy and the risk of post-ERCP pancreatitis. Surg Endosc. 2013 Jul;27(7):2498-503. doi: 10.1007/s00464-012-2768-4. Epub 2013 Jan 26. PMID 23355164
- [Result] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Result] Pan L, Chen M, Ji L, Zheng L, Yan P, Fang J, Zhang B, Cai X. The Safety and Efficacy of Laparoscopic Common Bile Duct Exploration Combined with Cholecystectomy for the Management of Cholecysto-choledocholithiasis: An Up-to-date Meta-analysis. Ann Surg. 2018 Aug;268(2):247-253. doi: 10.1097/SLA.0000000000002731. PMID 29533266
- [Result] Ricci C, Pagano N, Taffurelli G, Pacilio CA, Migliori M, Bazzoli F, Casadei R, Minni F. Comparison of Efficacy and Safety of 4 Combinations of Laparoscopic and Intraoperative Techniques for Management of Gallstone Disease With Biliary Duct Calculi: A Systematic Review and Network Meta-analysis. JAMA Surg. 2018 Jul 18;153(7):e181167. doi: 10.1001/jamasurg.2018.1167. Epub 2018 Jul 18. PMID 29847616
- [Result] Tan C, Ocampo O, Ong R, Tan KS. Comparison of one stage laparoscopic cholecystectomy combined with intra-operative endoscopic sphincterotomy versus two-stage pre-operative endoscopic sphincterotomy followed by laparoscopic cholecystectomy for the management of pre-operatively diagnosed patients with common bile duct stones: a meta-analysis. Surg Endosc. 2018 Feb;32(2):770-778. doi: 10.1007/s00464-017-5739-y. Epub 2017 Jul 21. PMID 28733744
- [Result] Tse F, Yuan Y, Moayyedi P, Leontiadis GI. Guide wire-assisted cannulation for the prevention of post-ERCP pancreatitis: a systematic review and meta-analysis. Endoscopy. 2013 Aug;45(8):605-18. doi: 10.1055/s-0032-1326640. Epub 2013 Jun 27. PMID 23807804
- [Result] Morino M, Baracchi F, Miglietta C, Furlan N, Ragona R, Garbarini A. Preoperative endoscopic sphincterotomy versus laparoendoscopic rendezvous in patients with gallbladder and bile duct stones. Ann Surg. 2006 Dec;244(6):889-93; discussion 893-6. doi: 10.1097/01.sla.0000246913.74870.fc. PMID 17122614
- [Result] Tatulli F, Cuttitta A. Laparoendoscopic approach to treatment of common bile duct stones. J Laparoendosc Adv Surg Tech A. 2000 Dec;10(6):315-7. doi: 10.1089/lap.2000.10.315. PMID 11132910